CLINICAL TRIAL: NCT05674422
Title: Circulating Tumor DNA as a Predictor of Relapse in Patients With Locally Advanced Rectal Cancer Treated With Total Neoadjuvant Therapy Followed by Watch and Wait or Total Mesorectal Excision Based on Clinical Assessment of Response
Brief Title: GEMCAD-REVEAL STUDY - Circulating Tumor DNA as a Predictor of Relapse in Patients With Locally Advanced Rectal Cancer.
Acronym: REVEAL
Status: Active, not recruiting | Type: Observational
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Responsible Party: Sponsor
Other Study IDs: GEMCAD 2201
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Patients With Locally Advanced Rectal Cancer
Keywords: rectal cancer; ctDNA; total neoadjuvant therapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA from liquid biopsy: he ctDNA isolation test selected for this study is marketed by Guardant Health (Redwood City, California, USA) under the name Guardant RevealTM. It consists of a single state-of-the-art liquid blood biopsy, which is capable of detecting residual or recurrent disease seven days after blood extraction. This test uses a sequencing method that simultaneously evaluates genetic alterations and methylation without the need for a biopsy of the primary tumor tissue to determine specific mutations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: total neoadjuvant therapy — All patients will be aged 18 years or older, with histologically confirmed rectal adenocarcinoma, located in the mid or distal third (with the inferior margin within 12cm from the anal verge), clinically staged II and III (cT3-T4 and/or any TN+), scheduled to undergo TNT will be eligible. All cases and treatment decisions will be discussed by local Multidisciplinary Boards

SUMMARY:
The evaluation of the tumor response to chemoradiotherapy/total neoadjuvant therapy (CRT/TNT) remains a challenge. The integration of a blood-based biomarker such as ctDNA with clinico-radiological tools could offer the potential advantage of improving accuracy of assessment of tumor response to neoadjuvant therapy. Furthermore, data on functional outcomes and quality of life after total mesorectal excision (TME) and especially after " Watch And Wait" (WW) is scarce.

REVEAL is a prospective, multicenter study in which the response to TNT in correlation with liquid biopsy (LB) of patients with rectal cancer in Spain will be evaluated. It is planned to include 120 patients. All patients will be aged 18 years or older, with histologically confirmed rectal adenocarcinoma, located in the mid or distal third (with the inferior margin within 12cm from the anal verge), clinically staged II and III (cT3-T4 and/or any TN+), scheduled to undergo TNT will be eligible. All cases and treatment decisions will be discussed by local Multidisciplinary Boards. Patients will be included consecutively when visiting the corresponding health centers for outpatient visits or hospitalization.

The objective of the present study is to evaluate the role of ctDNA in the prediction of relapse in patients diagnosed with locally advanced rectal cancer (LARC) treated with TNT followed by WW or TME based on a clinical assessment of the local response

DETAILED DESCRIPTION:
The evaluation of the tumor response to chemoradiotherapy/total neoadjuvant therapy (CRT/TNT) remains a challenge. The integration of a blood-based biomarker such as ctDNA with clinico-radiological tools could offer the potential advantage of improving accuracy of assessment of tumor response to neoadjuvant therapy. Furthermore, data on functional outcomes and quality of life after total mesorectal excision (TME) and especially after " Watch And Wait" (WW) is scarce.

REVEAL is a prospective, multicenter study in which the response to TNT in correlation with liquid biopsy (LB) of patients with rectal cancer in Spain will be evaluated. It is planned to include 120 patients. All patients will be aged 18 years or older, with histologically confirmed rectal adenocarcinoma, located in the mid or distal third (with the inferior margin within 12cm from the anal verge), clinically staged II and III (cT3-T4 and/or any TN+), scheduled to undergo TNT will be eligible. All cases and treatment decisions will be discussed by local Multidisciplinary Boards. Patients will be included consecutively when visiting the corresponding health centers for outpatient visits or hospitalization.

The objective of the present study is to evaluate the role of ctDNA in the prediction of relapse in patients diagnosed with locally advanced rectal cancer (LARC) treated with TNT followed by WW or TME based on a clinical assessment of the local response.

HYPOTHESIS ctDNA is a predictor of complete clinical response and could potentially be used to guide patient selection for WW strategy.

ctDNA is an early marker of local tumor relapse and could potentially guide strategy changes during follow-up.

Patients who are enrolled in a WW strategy have better long-term functional outcomes in comparison to patients who undergo surgery.

OBJECTIVES

PRIMARY:

To estimate the positive predictive value (PPV) and the negative predictive value (NPV) of the post-TNT ctDNA measurement to identify relapse (local or distant) in the 2 years after TNT.

SECONDARY:

Secondary objectives related to ctDNA and tumor response to TNT:

* To estimate the concordance between the post-TNT ctDNA measurement and the clinical evaluation of response (endoscopy-biopsy, DRE and MRI) to TNT.
* To estimate the concordance between the ctDNA measured after TNT and the endoscopy-biopsy evaluation of response.
* To estimate the concordance between the ctDNA measured after TNT and the MRI-defined response pattern groups.

Secondary objectives related to ctDNA measure during follow-up and relapse:

* To estimate the positive predictive value and the negative predictive value of ctDNA measured during the follow-up after TNT to identify relapse (local or distant) in the 2 years after TNT.
* To estimate the positive predictive value and the negative predictive value of ctDNA measured during the follow-up after TNT to identify local relapse in the 2 years after TNT
* To estimate the positive predictive value and the negative predictive value of ctDNA measured during the follow-up after TNT to identify distant relapse in the 2 years after TNT

Secondary objective related to functional impact of TME and WW:

-To describe anorectal, urinary and sexual function in the TME and WW groups.

Secondary objective related to ctDNA and survival:

-To assess the association of ctDNA levels (at baseline, post-treatment and during follow-up) with the survival outcomes (overall and disease-free survival, locoregional and distant recurrence, together with the pattern of recurrence).

ELIGIBILITY:
Inclusion Criteria:

* Legally capable patients ≥ 18 years of age.
* Histologically confirmed rectal adenocarcinoma.
* Any tumor located in the mid or distal rectum, clinically staged II-III (cT3/4 and/or any TN+).
* Willingness to be enrolled in the WW strategy if cCR or nCCR is achieved.
* Absence of metastases on imaging.
* Scheduled to undergo TNT followed by delayed surgery.
* Patients who have signed the informed consent for this study.

Note: Decision was taken to treat the patient with a specific treatment prior and independently of patient inclusion in this non interventional study.

Exclusion Criteria:

* Patients who do not meet inclusion criteria.
* Concomitant colorectal tumors.
* Intolerance or contraindication to planned TNT.
* Other concurrent malignant diseases. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with locally advanced rectal cancer candidates to TNT. All patients will be aged 18 years or older, with histologically confirmed rectal adenocarcinoma, located in the mid or distal third (with the inferior margin within 12cm from the anal verge), clinically staged II and III (cT3-T4 and/or any TN+), scheduled to undergo TNT will be eligible.
  All enrolled patients will be allocated to receive TNT according to standard clinical practice.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2025-04-26 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
ctDNA from liquid biopsy | 2 years after to start treatment total neoadjuvant therapy/2 years per patient
  The results from ctDNA will be dichotomized to positive or negative. The investigator will report the percentage of patients with positive or negative ctDNA. Correlation of these values with clinical endpoints of response / survival to total neoadjuvant therapy will be done to fulfill the proposed objectives of this study. The ctDNA isolation test selected for this study is marketed by Guardant Health (Redwood City, California, USA) under the name Guardant RevealTM. It consists of a single state-of-the-art liquid blood biopsy, which is capable of detecting residual or recurrent disease seven days after blood extraction. This test uses a sequencing method that simultaneously evaluates genetic alterations and methylation without the need for a biopsy of the primary tumor tissue to determine specific mutations.

SECONDARY OUTCOMES:
Response to TNT (cCR,nCCR) | Throughout the study period, approximately 2 years per patient
  Number of patients will be classified as responders (cCR, nCCR) or non responders based on the International Consensus Recommendations for Organ Preservation in Rectal Cancer. The number and percentage of each category will be reported.
  cCR: clinical complete response nCCR: near-complete clinical response
Response to TNT (WW or TME) | Throughout the study period, approximately 2 years per patient
  The number and percentage of patients allocated to "watch and wait" (WW) or Total Mesorectal Excision (TMT) will be provided. Response rates will be also provided separately depending on the technique empowered to determine the response:
  * Endoscopy-biopsy
  * MRI
Locoregional failure rate (LRF) | Throughout the study period, approximately 2 years per patient
  Locoregional failure rate (LRF) defined as the percentage of patients who present progression(only for patients with nCCR)/relapse of disease in the rectum, regional organs and/or regional lymph nodes. Locoregional failure rate will be estimated using the appropriate logistic regression model at 1-year after the first dose of TNT and end of study. Those patients lost to follow-up with no event of local recurrence will be considered not evaluable for LFR endpoint. Patients who die as a direct or secondary cause of the cancer will be considered as an event at the date of death for LFR analysis. Death by other reasons other than cancer progression/relapse will not be considered as an event for LFR.
Distant relapse rate (DRR) | Throughout the study period, approximately 2 years per patient
  Distant relapse rate (DRR) defined as the percentage of patients who present progression/relapse of disease in distant locations. DRR will be estimated using the appropriate logistic regression model at 1-year after the first dose of TNT and end of study. Those patients lost to follow-up with no event of distal recurrence will be considered not evaluable for DRR endpoint. Patients who die as a direct or secondary cause of the cancer will be considered as an event at the date of death for DRR analysis. Death by other reasons other than cancer progression/relapse will not be considered as an event for DRR.
Disease-free Survival (DFS) | at 1 year after the first dose of TNT and at the end of study (approximately 2 years)
  Disease-free Survival (DFS): defined as the time elapsed from the first dose of TNT to progression (only for pts with nCCR), relapse, or death from any cause, whichever occurs first. The investigators will assess the median DFS, the DFS rate at 1 year, and at the end of study. The 1-year DFS rate is defined as the rate of patients alive and free of relapse or progression at 1 year after the first dose of TNT estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment.
Disease-specific Survival (DSS) | at 1 year after the first dose of TNT
  Disease-specific Survival (DSS): defined as the time elapsed from the first dose of TNT to the date of progression(only for pts with nCCR), relapse, or death due to the disease, whichever occurs first. We will assess the median DSS, the DSS rate at 1 year, and at the end of study. The 1-year DSS rate is defined as the rate of patients alive and free of event at 1 year after the first dose of TNT, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Overall Survival (OS) | at 1 year after the first dose of TNT
  Overall Survival (OS) : defined as the time elapsed from the first dose of TNT until death from any cause. We will assess the median OS and the OS rate at 1 year. The 1-year OS rate is defined as the rate of patients alive at 1 year after the first dose of TNT, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Mortality | Throughout the study period, approximately 2 years per patient
  Mortality: Rate of patients who died during the study. The number and percentage of patients will be provided.
TNT compliance | Throughout the study period, approximately 2 years per patient
  TNT compliance: total number of dose reductions and modifications of the treatment throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Yoelimar Guzmán, M.D., Study Chair — Servicio de Cirugía General y Digestiva, Hospital Clínic, Universitat de Barcelona; Joan Maurel Santasusana, M.D., Ph.D., Study Chair — Servicio de Oncología, Hospital Clínic, Universitat de Barcelona; Juan Ramón Ayuso, M.D., Ph.D., Study Chair — Servicio de Radiología, Hospital Clínic, Universitat de Barcelona
Locations (15):
- Spain (15):
  - Hospital Germans Trias i Pujol - ICO Badalona, Badalona, Barcelona
  - Hospital Universitari Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - H. de la Santa Creu i Sant Pau, Barcelona
  - H.U. Vall d'Hebron, Barcelona
  - Hospital Clínic, Universitat de Barcelona, Barcelona
  - Hospital Del Mar, Barcelona, Barcelona
  - Hospital Sant Joan Despí - Moisés Broggi., Barcelona
  - ICO-Hospitalet, Barcelona
  - ICO Girona, Girona
  - H. Univeristario La Paz, Madrid
  - Hospital Quirón Salud Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No